CLINICAL TRIAL: NCT05628272
Title: Clinical Study of Cord Blood MNCs in the Treatment of Bone Marrow Failure After Chemotherapy in Children With Malignant Diseases
Brief Title: MNCs for Bone Marrow Failure After Malignant Diseases Children Chemotherapy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Qianfoshan Hospital (Other)
Collaborators: Chinese Medical Association (Network)
Responsible Party: Principal Investigator, Gu Yan, professor, Qianfoshan Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SDDYYK-KY0913
Record Dates: First submitted 2022-09-15; First posted 2022-11-28 (Actual); Last update posted 2022-11-28 (Actual); Status verified 2022-11

CONDITIONS: Cord
Keywords: bone marrow failure; pediatric chemotherapy; mononuclear cells
MeSH Terms: conditions — Cone-Rod Dystrophies; Bone Marrow Failure Disorders

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): granulocyte stimulating factor(5ug/kg/d) +infusion of umbilical cord blood mononuclear cells, each infusion ≥1×10^8, once a week
  Interventions: Other: Intravenous infusion of cord blood mononuclear cells; Drug: application of granulocyte stimulating factor
- control group (Placebo Comparator): granulocyte stimulating factor 5ug/kg/d
  Interventions: Drug: application of granulocyte stimulating factor

INTERVENTIONS:
Other: Intravenous infusion of cord blood mononuclear cells — On the basis of the application of granulocyte stimulating factor, the research group was given intravenous infusion of umbilical cord blood mononuclear cells, each infusion ≥1×10^8, once a week
  Arms: Experimental group
Drug: application of granulocyte stimulating factor — application of granulocyte stimulating factor

SUMMARY:
This project aims to investigate the therapeutic and repair effects of cord blood mononuclear cells (MNCs) on bone marrow failure after chemotherapy in children with malignant diseases. It is planned to collect 20 malignant children with bone marrow failure after chemotherapy and randomly divide them into two groups. The umbilical cord blood mononuclear cells were injected, ≥1×10^8 per infusion, once a week, and the recovery time of peripheral blood leukocytes, neutrophils, platelets and hemoglobin was observed. According to the recovery of myelosuppression, stop when the peripheral blood reaches leukocytes>1×10^9/L, neutrophils>0.5×10^9/L, platelets>25×10^9/L, and hemoglobin>60g/L at the same time. Use, share 1-4 times.

Statistical software was used to compare the changes of peripheral blood leukocytes, neutrophils, platelets and hemoglobin before the start of the test (0d) and 1d, 3d, 5d, 7d, 10d, and 14d after the start of the test, as well as the severity of concurrent infections and antibiotic use Time, number of infusions of blood products.

DETAILED DESCRIPTION:
The standard of bone marrow failure after chemotherapy is based on theWorld Health Organization(WHO) grade IV myelosuppression standard, that is, peripheral blood white blood cells (WBC) < 1 × 10^9/L, neutrophils (N) <0.5 × 10^9/L, platelets (PLT) <25×10^9/L, hemoglobin (Hb) <60g/L, for more than 2 weeks. It is planned to collect 20 malignant children with bone marrow failure after chemotherapy and randomly divide them into two groups. The umbilical cord blood mononuclear cells were injected, ≥1×10^8 per infusion, once a week, and the recovery time of peripheral blood leukocytes, neutrophils, platelets and hemoglobin was observed. According to the recovery of myelosuppression, when the peripheral blood reaches WBC>1×10^9/L, N>0.5×10^9/L, PLT>25×10^9/L, and Hb>60g/L at the same time, it should be discontinued and used together. 1-4 times.

Safety evaluation: Children under treatment who meet any one or more of the following, the study will be terminated or withdrawn: (1) Within 6 hours after the treatment with venous cord blood mononuclear cells, the clinical symptoms that cannot be explained by known causes are significantly aggravated or In case of deterioration, the trial should be terminated, and appropriate treatment should be carried out. The withdrawn cases should be included in the clinical efficacy evaluation, and the count is invalid; (2) During the treatment and within 6 hours after the treatment, the following conditions that cannot be explained by the known causes occur: severe hypotension, contraction Blood pressure drops ≥20mmHg or systolic blood pressure <70mmHg; severe hypertension, systolic blood pressure rises ≥20mmHg or systolic blood pressure>140mmHg, the test should be terminated; (3) During treatment and within 6 hours after treatment, chills, Patients with fever (body temperature ≥39°C), rash, headache, low back pain and other symptoms should stop the test; (4) If serious adverse events occur, the test should be stopped.

Efficacy evaluation: compare the changes of peripheral blood leukocytes, neutrophils, platelets and hemoglobin before the start of the test (0d) and 1d, 3d, 5d, 7d, 10d, and 14d after the start of the test, as well as the severity of concurrent infection and antibiotic use Time, number of infusions of blood products.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≤ 17 years old;
2. Treated in pediatric hematology department from September 2021 to September 2024, patients with bone marrow failure after transplantation;
3. Eastern Cooperative Oncology Group(ECOG) score ≤ 2;
4. Sign the informed consent form (< 10 years old, signed by the guardian; ≥ 10 The children and their guardians signed the informed consent form before the selection.

Exclusion Criteria:

1. Those who have received thoracic radiotherapy in the past;
2. Those who do not meet the above inclusion criteria.

Ages: 1 Year to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Estimated)
Dates: Start 2022-10-01 (Actual); Primary Completion 2024-09-01 (Estimated); Study Completion 2024-09-01 (Estimated)

PRIMARY OUTCOMES:
recovery time of peripheral neutrophils | 20days
  Observe the recovery time of peripheral neutrophils

SECONDARY OUTCOMES:
frequency of infection | 20days
  frequency of infection

CONTACTS AND LOCATIONS:
Overall Officials: Yan GU, Professor, Study Director — Qianfoshan Hospital
Locations (1):
- Pediatrics, Qianfoshan Hospital, Jinan, Shandong, China

IPD SHARING:
Plan to Share IPD: No
To be published in an appropriate form at the complete conclusion of the study